CLINICAL TRIAL: NCT07172581
Title: Impact of an Online Service Offering Personalized Low-FODMAP Menus With Nutritional Support on Quality of Life and Control of Physical and Psychological Symptoms in People With Irritable Bowel Syndrome
Brief Title: Online Low-FODMAP Diet in Irritable Bowel Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 19.304
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Online low-FODMAP diet (Experimental): An innovative approach was developed by the SOSCuisine® platform, an online menu service adapted to different conditions, including IBS. It enables people living with IBS to follow the FODMAP protocol in a self-service context, using online resources of personalized weekly low-FODMAP menus, instructions for each phase and a peer support group moderated by a specialized registered dietitian.
  Interventions: Behavioral: Online low-FODMAP diet

INTERVENTIONS:
Behavioral: Online low-FODMAP diet — Participants were invited to follow the online low-FODMAP diet offered by SOSCuisine®, characterized by three specific features. First, participants received customized weekly low-FODMAP menus based on the Monash University protocol. Second, a virtual assistant accompanied participants from the beginning to the end of the diet implementation, providing personalized recommendations tailored to individual's preferences and intensity of symptoms. For the reintroduction phase, the assistant guided individuals through the process of testing specific FODMAP subgroups, offering food suggestions based on individual preferences, and portion sizes. The last feature of the platform was the access to a peer support group on Facebook©, designed to foster communication among participants. This group allowed individuals to ask questions and receive valid answers, as the group was moderated by a FODMAP-specialized registered dietitian.

SUMMARY:
This study aimed to assess the impact of implementing the low Fermentable Oligo-, Di- and Monosaccharides, And Polyols (FODMAP) diet, through an online educational service platform, on the quality of life of patients living with irritable bowel syndrome (IBS). A prospective single-group intervention pilot study involving patients with IBS from two hospitals was conducted. Participants followed the low FODMAP diet using a web-based platform for 6 months. The IBS quality of life questionnaire (IBS-QoL), the IBS symptom severity scoring system (IBS-SSS) and the State-Trait Anxiety Inventory Form Y (STAI) were completed at baseline, after the restriction phase and after reintroduction phase.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of IBS according to the Rome IV criteria by a gastroenterologist within the past three months
* understand French
* have an Internet access and a Facebook© account with a self-reported familiarity to use them

Exclusion Criteria:

* patients suffering from a known eating or mental health disorder
* body mass index under 18.5 kg/m2
* type 1 or 2 diabetes
* pregnancy
* other chronic gastrointestinal diseases, except gastroesophageal reflux

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-05-23 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
IBS-related quality of life | From enrollment to the end of intervention at 6 months.
  The primary outcome was the change in QoL from baseline to the end of study, assessed by the validated IBS-QoL questionnaire. This questionnaire assesses 8 domains, namely dysphoria, interference with activity, body image, health worry, food avoidance, social reaction, sexual concerns and relationships, from which a computed score is drawn. This score, ranging from 0 to 100, was developed to assess the self-reported QoL in IBS, a higher score indicating a better QoL.

SECONDARY OUTCOMES:
Severity of IBS symptoms | From enrollment to the end of intervention at 6 months.
  Secondary outcomes included changes in severity of IBS symptoms, measured by the validated IBS-Severity Scoring System (IBS-SSS). This questionnaire evaluates 5 specific domains within the last ten days: abdominal pain severity, abdominal pain duration, abdominal distension, bowel habits dissatisfaction and interference with life. A composite score is calculated and varies from 0 to 500. Depending on the score, the severity can be classified in 4 categories: absence of symptoms severity or remission (score < 75), mild (score 75-174), moderate (score 175-299), and severe (score ≥ 300).
State and trait anxiety | From enrollement to the end of intervention at 6 months.
  Anxiety was evaluated by the French-Canadian adaptation of the State-Trait Anxiety Inventory Form Y (STAI), which specifically assesses state anxiety (STAI-S), the subjective and transient emotional state of anxiety, and trait anxiety (STAI-T), a more stable predisposition to anxiety. The STAI-S score can be classified in 5 categories: very low state anxiety (score < 36), low (score 36-45), moderate (score 46-55), high (score 56-65), and very high (score > 65). For the STAI-T score, a score inferior to 40 commonly indicates low trait anxiety while a score of 40 or more indicates high trait anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de recherche du Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No